CLINICAL TRIAL: NCT00620048
Title: Injection of Autologous CD34+ Cells for Neovascularization and Symptom Relief in Patients With Myocardial Ischemia and LVEF < 40%
Brief Title: Stem Cell Study for Subjects With Congestive Heart Failure
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to lack of funding.
Sponsor: Losordo, Douglas, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00002516; 11196-03 (Other: Sponsor protocol number)
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2011-11

CONDITIONS: Myocardial Ischemia; Congestive Heart Failure; Cardiovascular Disease
Keywords: heart; stem Cells; low EF; heart attack; cardiomyopathy; congestive heart failure; cardiovascular disease; Heart Failure; Low Ejection Fraction
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure; Cardiovascular Diseases; Myocardial Infarction; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose of autologous CD34-positive cells (stem cells) (Experimental)
  Interventions: Biological: Intramyocardial injection of autologous CD34-positive cells (stem cells)
- High dose of autologous CD34-positive cells (stem cells) (Experimental)
  Interventions: Biological: Intramyocardial injection of autologous CD34-positive cells (stem cells)

INTERVENTIONS:
Biological: Intramyocardial injection of autologous CD34-positive cells (stem cells) — Comparison between a low dose and high dose of autologous (one's own) CD34-positive cells (stem cells) delivered via injections into the heart muscle.

SUMMARY:
The purpose of this study is to determine if cell therapy with your own cells (autologous cells) delivered with a catheter to regions of the heart with poor blood flow will be safe and if it will improve your ejection fraction and heart failure symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 21 to 80 years old (inclusive).
* Subjects with functional class (NYHA) II or III ischemic heart failure.
* Subjects who have attempted "best" cardiac medical therapy including long-acting nitrates, maximal use of beta-adrenergic blocking agents, and angiotensin-converting enzyme (ACE)inhibitors without control of symptoms.
* Subjects must be identified as non-candidates for conventional revascularization by their referring cardiologist.
* Subjects must have left ventricular ejection fraction <40% by echocardiography.
* All subjects must have a recent coronary angiogram (within the last 6 months) to document the coronary anatomy and insure the presence of coronary disease that is not amenable to standard revascularization procedures.
* Have serum B-type Natriuretic Peptide (BNP) level >100 pg/ml.

Exclusion Criteria:

* Myocardial infarction (Q wave or non-Q wave defined as CKMB >3 times normal) within 30 days of treatment.
* Successful coronary revascularization procedures within 3 months of study enrollment.
* Documented stroke or transient ischemic attack (TIA) within 60 days of study enrollment.
* NYHA Class IV heart failure and patients with idiopathic or non-ischemic heart failure.
* History of severe aortic stenosis (aortic valve area < 1.0 cm2) or insufficiency (>2+); severe mitral stenosis (mitral valve area <1.5 cm2); or severe mitral insufficiency(>2+).
* Implantation of biventricular pacemaker within 90 days of study treatment.
* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year, such as chronic medical illness (i.e. severe chronic obstructive pulmonary disease, renal failure or cancer).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety of intramyocardial administration of CD34-positive cells | 6 months

SECONDARY OUTCOMES:
Effects of intramyocardial injections of autologous CD34-positive cells on clinical outcomes. | 6 months
  Clinical outcomes assessed include symptoms, change in health status, myocardial function and exercise duration.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Losordo, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States